CLINICAL TRIAL: NCT03457896
Title: A Phase II Study Evaluating the Combination of Neratinib Plus Trastuzumab or Neratinib Plus Cetuximab in Patients With "Quadruple Wild-Type" (KRAS/NRAS/BRAF/PIK3CA Wild-Type) Metastatic Colorectal Cancer Based on HER2 Status: Amplified, Non-Amplified (Wild-Type) or Mutated
Brief Title: Study of Neratinib +Trastuzumab or Neratinib + Cetuximab in Patients With KRAS/NRAS/BRAF/PIK3CA Wild-Type Metastatic Colorectal Cancer by HER2 Status
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FC-11
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: NSABP; PUMA; Neratinib; Trastuzumab; Cetuximab; RAS; NRAS; BRAF; PIK3CA wild-type; Quadruple wild-type; HER2 status
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trastuzumab; Cetuximab; neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Experimental): Guardant360 test on blood from select patients with known HER2 status.
  Prior to assignment to Arm 1, HER2 test on blood obtained from Quadruple Wild-Type patients who received anti-EGFR therapy. Patients with HER2 amplified, HER2 Wild-Type or HER2 mutated will recieve:
  • Neratinib daily + Trastuzumab weekly until disease progression
  Interventions: Drug: Trastuzumab; Drug: Neratinib; Diagnostic Test: Guardant360 Diagnostic Test
- Arm 2 (Experimental): Patients with HER2 Wild Type or HER2 amplified with no prior anti-EGFR therapy will receive:
  • Neratinib daily + Cetuximab weekly until disease progression
  Interventions: Drug: Cetuximab; Drug: Neratinib

INTERVENTIONS:
Drug: Trastuzumab — Patients with HER2 amplified tumors with prior anti-EGFR therapy and/or HER2 mutated colorectal cancer with/or without prior anti-EGFR therapy will receive 4 mg/kg IV loading dose; then 2 mg/kg IV weekly until disease progression. Neratinib: 240 mg taken by mouth daily until disease progression.
  Arms: Arm 1
Drug: Cetuximab — Patients with HER2 WT or HER2 amplified with no prior anti-EGFR therapy: 400 mg/m2 IV loading dose; then 250 mg/m2 IV weekly. Neratinib 240 mg taken by mouth daily until disease progression.
  Arms: Arm 2
Drug: Neratinib — 240 mg taken by mouth daily until disease progression.
  Other Names: Nerlynx
Diagnostic Test: Guardant360 Diagnostic Test — Prior to assignment to Arm 1, the Guardant360 diagnostic test will be conducted in blood to confirm known HER2 status for select patients.
  Arms: Arm 1

SUMMARY:
This is a phase II trial to examine the efficacy of neratinib plus trastuzumab or neratinib plus cetuximab in patients with "quadruple wild-type" (all RAS/NRAS/BRAF/PIK3CA wild-type), metastatic colorectal cancer based on HER2 status (amplified, non-amplified [wild-type] or mutated). Patients must have confirmed quadruple wild-type (WT) genotype, via NSABP MPR-1 or from colonic biopsy or a metastatic biopsy taken prior to treatment, and known HER2 status.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the progression-free survival (PFS) in each of these HER2 populations. Secondary aims include overall response rate (ORR) and clinical benefit rate (CBR) defined as the objective tumor decrease and stable disease by RECIST 1.1 criteria; toxicity and safety profile. Exploratory analysis will be performed to assess for molecular predictors of response. The local site will make the primary determination of response and progression based on all radiographic images (e.g., MRI, CT, PET, bone scan, etc.) as well as other relevant reports documenting disease response or progression.

For patients identified as quadruple WT with prior cetuximab or panitumumab treatment, a pre-entry blood sample will be required from consenting patients to confirm HER2 amplification for study eligibility.

Patients with quadruple WT, HER2 amplified with prior anti-EGRF therapy and/or HER2 mutated colorectal cancer with/or without prior anti-EGRF therapy will receive concurrent therapy with trastuzumab 4 mg/kg IV loading dose followed by 2 mg/kg IV weekly and neratinib 240 mg taken by mouth daily until disease progression, (Arm 1).

Patients with quadruple WT, HER2 WT or HER2 amplified with no prior anti-EGRF therapy will be assigned to receive concurrent therapy with cetuximab (400 mg/m2 IV loading dose followed by 250 mg/m2 IV weekly), and neratinib 240 mg taken by mouth daily until disease progression (Arm 2).

Approximately thirty-five (35) patients will be accrued to this study; 15 patients with HER2 amplified, 15 patients with HER2 WT, and approximately 5 patients with HER2 mutated colorectal cancer. Patients with HER2 WT or HER2 amplified mCRC who drop out of the study before the first scan (for whatever reason) will be replaced. Patients who drop out of the study after the first scan but before the second scan will be considered to have progressive disease.

Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).

Required blood and tissue samples will be collected at entry into the study. A tumor biopsy will be procured from an accessible site of metastasis before study therapy is initiated (after the patient has signed the consent form and has been screened for eligibility). Tissue will be sent to Champions Oncology Laboratory for engraftment into an NOD/SCID mouse to develop a patient-derived xenograft (PDX) model, and to NSABP Pathology Division for correlative science. Tissue samples from PDX models will be sent to Celcuity for functional HER2 signaling assay. Additional blood samples will be collected during the course of treatment.

Optional tumor and blood samples will be collected from consenting patients at the time of disease progression.

ELIGIBILITY:
Inclusion Criteria:

The tumor tissue must have been determined to be KRAS, NRAS, BRAF, PIK3CA (all RAS quadruple) wild-type by CLIA testing.

The ECOG performance status must be 0, 1 or 2. Patients must have the ability to swallow and retain oral medication. There must be documentation by CT scan, or MRI, that the patient has evidence of measurable metastatic disease per RECIST 1.1 criteria.

Patients must have an accessible metastatic lesion for pretreatment core biopsy procurement.

Unless either drug is medically contraindicated, patients must have received oxaliplatin and irinotecan as part of standard chemotherapy regimens. (This includes adjuvant therapy.)

Specific patient eligibility for quadruple WT and HER2 status:

Arm 1:

HER2 amplified confirmed by CLIA testing performed on blood samples, and prior treatment with cetuximab or panitumumab.

HER2 mutation confirmed by CLIA testing of tumor, and with or without prior treatment with cetuximab or panitumumab.

Arm 2:

HER2 WT or HER2 amplified confirmed by CLIA testing of this tumor, and no prior therapy with cetuximab or panitumumab.

Blood counts performed within 2 weeks prior to study entry must meet the following criteria:

ANC must be greater than or equal to 1000/mm3. Platelet count must be greater than or equal to 75,000/mm3. Hemoglobin must be greater than or equal to 8 g/dL.

Adequate hepatic function performed within 2 weeks prior to study entry must be met:

* Total bilirubin must be less than or equal to 1.5 x ULN (upper limit of normal) for the lab unless the patient has a bilirubin elevation greater than 1.5 x ULN to 3 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
* Alkaline phosphatase must be less than or equal to 3 x ULN for the lab with the following exception: for patients with documented liver metastases or bone involvement alkaline phosphatase must be less than or equal to 5 x ULN; and
* AST and ALT must be less than or equal to 3 x ULN for the lab with the following exception: for patients with documented liver metastases, AST and ALT must be less than or equal to 5 x ULN.

Serum creatinine performed within 2 weeks prior to study entry must be less than or equal to 1.5 x ULN for the lab.

Patients eligible for Arm 1 (neratinib + trastuzumab): Left ventricular ejection fraction must be greater than or equal to 50% or within normal range for the institution (whichever is lowest).

Female patients and male patients with female partners of reproductive potential must agree to use an effective method of contraception during therapy and for at least 7 months after the last dose of study therapy.

Exclusion Criteria:

Diagnosis of anal or small bowel carcinoma. Colorectal cancer histology other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.

Previous therapy with any HER2 targeting agents (such as trastuzumab, lapatinib, neratinib, etc.) for any malignancy.

Symptomatic brain metastases or brain metastases requiring chronic steroids to control symptoms.

Active hepatitis B or hepatitis C with abnormal liver function tests. Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function.

Persistent CTCAE v4.0 greater than or equal to grade 2 diarrhea regardless of etiology.

CTCAE v4.0 grade 3 or 4 anorexia or nausea related to metastatic disease. CTCAE v4.0 greater than or equal to grade 2 vomiting related to metastatic disease.

Any of the following cardiac conditions: documented congestive heart failure; myocardial infarction within 6 months prior to study entry; unstable angina within 6 months prior to study entry; symptomatic arrhythmia.

Serious or non-healing wound, skin ulcer, or bone fracture. History of bleeding diathesis. (Patients on stable anticoagulant therapy are eligible.) Symptomatic interstitial lung disease or definitive evidence of interstitial lung disease described on CT scan, MRI, or chest x-ray in asymptomatic patients; dyspnea at rest requiring current continuous oxygen therapy.

Previous serious hypersensitivity reaction to monoclonal antibodies. (Determination of "serious" hypersensitivity reaction is at the investigator's discretion.) Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy greater than or equal to 12 months prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, colorectal carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing should be performed within 14 days prior to study entry according to institutional standards for women of childbearing potential.) Use of any investigational agent within 4 weeks prior to study entry. Note: Use of agents known to be strong cytochrome P450 (CYP) 3A4 inducers or inhibitors, and proton pump inhibitors (PPIs) should be avoided for the duration of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival with neratinib plus trastuzumab therapy | From initiation of neratinib plus trastuzumab therapy to time of tumor assessment, between cycle 6 and 7,which is usually six months after start of therapy.
  Progression free survival (PFS). Percentage of patients alive with absence of progression assessed using RECIST 1.1 criteria.
Progression free survival (PFS) with neratinib plus cetuximab therapy | From initiation of neratinib plus cetuximab therapy to time of tumor assessment between cycles 6 and 7, which is usually 6 months after start of therapy
  Progression free survival (PFS). Percentage of patients alive with absence of progression assessed using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall response rate to study therapy | From initiation of study therapy until disease progression, approximately 6 months.
  Rate of best overall response using measurement of tumor in patients with measurable metastatic disease
Clinical benefit rate | From initiation of study therapy until disease progression, approximately 6 months.
  Rate of disease status by continuous tumor measurement.
Frequency of adverse events assessed using CTCAE 4.0 | From beginning of study therapy until disease progression, approximately 6 months.
  Frequency of adverse events categorized using the NCI Common Terminology Criteria for Adverse Events version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (48):
- United States (48):
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente-Sunset, Los Angeles, California
  - Kaiser Permanente-West Los Angeles (Cadillac), Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-Sacramento, Sacramento, California
  - Kaiser Permanente-Medical Group, San Diego, California
  - Kaiser Permanente-Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-San Jose, San Jose, California
  - Kaiser Permanente-San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente Medical Center Santa Clara, Santa Clara, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UF Health Davis Cancer Pavilion and Shands Medical Plaza, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Cancer Care Specialists of Central IL-Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crosslands Cancer Center, Effingham, Illinois
  - Cancer Care Specialists of Central IL-Swansea, Swansea, Illinois
  - Trinity Health Michigan, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - St. Joseph Mercy Brighton, Brighton, Michigan
  - St. Joseph Mercy Canton, Canton, Michigan
  - St. Joseph Mercy Chelsea, Chelsea, Michigan
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - Spectrum Health Butterworth, Grand Rapids, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - St. Mary's of Michigan, Saginaw, Michigan
  - Lakeland Healthcare-Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Minnesota Oncology-Fridley, Saint Louis Park, Minnesota
  - Thomas Jefferson University Hospital-Sidney Kimmel Cancer Network, Philadelphia, Pennsylvania
  - Wellmont Cancer Institute, Johnson City, Tennessee
  - Wellmont Cancer Institute, Kingston, Tennessee
  - Wellmont Medical Associates-Oncology and Hematology, Bristol, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia

REFERENCES:
- [Derived] Freeman TJ, George TJ, Jacobs SA, Yothers G, Kolevska T, Feng H, Lipchik C, Maley S, Song N, Srinivasan A, Finnigan M, Wade JL 3rd, Buchschacher GL Jr, Al Baghdadi T, Shipstone A, Lin D, Puhalla SL, Allegra CJ, Wolmark N, Pogue-Geile KL. NSABP FC-11: A phase II study of neratinib plus trastuzumab or neratinib plus cetuximab in patients with "quadruple wild-type" (KRAS/NRAS/BRAF/PIK3CA) metastatic colorectal cancer based on HER2 status: amplified, non-amplified (wild-type), or mutated. Cancer Chemother Pharmacol. 2025 Aug 9;95(1):80. doi: 10.1007/s00280-025-04802-8. PMID 40782152